CLINICAL TRIAL: NCT00142883
Title: The Effects of GABA Medications on Cocaine Responses in Humans
Brief Title: The Effects of GABA Enhancing Medications on Individuals Addicted to Cocaine - 3
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has been completed
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Principle Investigator, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-18197-3; P50DA018197-03 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Cocaine Abuse; Cocaine-Related Disorders
Keywords: addiction, crack, cocaine
MeSH Terms: conditions — Cocaine-Related Disorders; Behavior, Addictive | interventions — Pregabalin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pregabalin (Active Comparator): pregabalin compared to placebo
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Placebo compared to pregabalin
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Pregabalin — pregabalin compared to placebo
  Other Names: lyrica
  Arms: pregabalin
Drug: placebo — sugar pill compared to pregabalin
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
Gamma-aminobutyric acid (GABA) is a type of neurotransmitter, which is a chemical that transmits information within and from the brain to all parts of the body. By lowering the level of another neurotransmitter called dopamine, GABA may have the ability to diminish cocaine cravings in addicts. The purpose of this study is to gather information on the interaction between cocaine and selected GABA enhancing medications in individuals addicted to cocaine. This may lead to future clinical studies using GABA medications to treat cocaine addiction.

DETAILED DESCRIPTION:
GABA is an inhibitory neurotransmitter that is found primarily in the brain. High GABA levels result in low levels of dopamine, another neurotransmitter that is the brain's "feel good" chemical and which plays a primary role in cocaine drug addiction. Cravings for cocaine can be reduced by lowering dopamine levels. This makes GABA-altering medications a potential treatment for cocaine addiction. This study will involve five GABA enhancing medications: tiagabine, topiramate, valproic acid, baclofen, and progesterone. The purpose of the study is to evaluate the interaction between GABA medications and cocaine in terms of safety and craving responses. In turn, these findings may guide future cocaine pharmacotherapy trials.

This 6-day inpatient study will begin with an orientation session to familiarize participants with study procedures. The evening of Day 1, all participants will receive placebo medication. On Days 2 through 4, participants will receive one of five GABA medications. The GABA medications will be given in gradually increasing doses to attain therapeutic levels while maintaining safety and minimizing side effects. Three experimental cocaine sessions will take place; one while the participants are receiving the placebo medication and two while the participants are receiving the GABA medications. During these sessions, cocaine will be administered intravenously in three increasing doses, each separated by 30-minute intervals. This will allow the participants' subjective and physiological responses during cocaine administration to return to baseline levels before the next dose. Blood will be drawn after each dose; heart rate, blood pressure, and an ECG will be monitored throughout the sessions. At the end of each session, questionnaires will be administered to assess the effects of cocaine and related mood states, as well as allow the participants to report any adverse events, depression, craving, or withdrawal symptoms.

This study is now closed and published.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for cocaine dependence
* History of smoked or intravenous cocaine use on average of at least once a week over a 6 month period
* Positive urine test for cocaine
* No current medical problems
* Normal electrocardiogram
* If female, willing to use contraception throughout the study

Exclusion Criteria:

* Seeking treatment for cocaine dependence
* Current major psychiatric illness, including mood disorder, psychotic disorder, or anxiety disorder
* Current dependence on alcohol or any drugs other than cocaine or nicotine
* History of major medical illness, including liver disease, suspected or known cancer, thrombophlebitis, or other medical conditions that are considered unsafe for study participants by the investigator
* Known allergy to study medications
* Pregnant or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2004-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Analog rating scale for drug effects; measured during each experimental session | one week
Physiological response to cocaine; measured during each experimental session | one week

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Kosten, MD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States